CLINICAL TRIAL: NCT02523079
Title: Cognitive Behavioral Therapy for Insomnia Among Different Types of Shift Workers
Acronym: CBT-INSOMNIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: Finnish Work Environment Fund (Other); NordForsk (Unknown); City of Helsinki (Other); City of Turku, Occupational Health Centre (Unknown); Finnair Health Services (Unknown); Aava Medical Centre (Other); Fazer Health Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34627; 114391 (Other Grant/Funding Number: Finnish Work Environment Fund); 53/13/03/00/15 (Registry Identifier: The Ethics Committees of the Hospital District of Helsinki and Uusimaa, Finland); 74809 (Other Grant/Funding Number: NordForsk)
Record Dates: First submitted 2015-07-01; First posted 2015-08-14 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Insomnia; Cognitive Behavioral Therapy; Sleep Disorders, Circadian Rhythm; Sleep Disorders, Shift-Work
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Behavioral Group Therapy for Insomnia (Experimental): Includes 6 group sessions (90 minutes each). The groups are led by trained psychologist or nurse of occupational health services. The manualized treatment is based on the general CBT-I model and includes components such as sleep hygiene, relaxation, stimulus control, sleep restriction and cognitive restructuring. In addition, participants receive information on how to schedule sleep, wake and light based on circadian principles while working differently timed shifts.
  Interventions: Behavioral: Cognitive Behavioral Group Therapy for Insomnia
- Cognitive Behavioral Self-help Therapy for Insomnia (Experimental): Mainly computerized self-help intervention. Includes an individual session before and after the intervention (30 minutes each) led by trained psychologist or nurse of occupational health services. The self-help treatment is based on the general CBT-I model and includes components such as sleep hygiene, relaxation, stimulus control, sleep restriction and cognitive restructuring. In addition, participants receive information on how to schedule sleep, wake and light based on circadian principles while working differently timed shifts.
  Interventions: Behavioral: Cognitive Behavioral Self-help Therapy for Insomnia
- Sleep Hygiene Guidance (Experimental): Includes one individual session (60 minutes) led by trained psychologist or nurse of occupational health services. The intervention is based on sleep hygiene guidance.
  Interventions: Behavioral: Sleep Hygiene Guidance

INTERVENTIONS:
Behavioral: Cognitive Behavioral Group Therapy for Insomnia
  Other Names: Group-based CBT-I
  Arms: Cognitive Behavioral Group Therapy for Insomnia
Behavioral: Cognitive Behavioral Self-help Therapy for Insomnia
  Other Names: Self-help CBT-I
  Arms: Cognitive Behavioral Self-help Therapy for Insomnia
Behavioral: Sleep Hygiene Guidance
  Arms: Sleep Hygiene Guidance

SUMMARY:
The aim of the study is to compare the implementation and effectiveness of group and self-help based cognitive behavioral treatment for insomnia (CBT-I) delivered by occupational health services (OHS) in a randomized and controlled design (RCT) among different types of shift workers.

DETAILED DESCRIPTION:
Because of irregular sleep-wake pattern shift work is a challenge in the screening and treatment of chronic insomnia. Earlier results has showed that CBT-I delivered by trained nurses of OHS may be effective treatment also among workers with irregular work hours. The aim of the present study is to compare the implementation and effectiveness of OHS delivered group and self-help based CBT-I in a RCT design among different types of shift work.

Participants (n=90-120) are shift workers with insomnia disorder that has lasted at least three months. The participants are randomized to a) group-based CBT-I (6 group sessions); or b) mainly computerized self-help CBT-I (an individual session before and after the intervention) delivered by a trained OHS nurse or psychologist; or c) control group given a sleep hygiene intervention (1 individual session). Outcomes are assessed using a sleep diary, questionnaires, actigraphy and cognitive performance tests. To study the effect of CBT-I program at molecular level, blood samples of participants will be collected at baseline and at the end of the program for genetic analyses. The measurements are conducted at five time points for a period of two years.

The investigators expect to find that both group and self-help based CBT-I among different types of shift workers are effective low-intensity treatments of chronic insomnia compared to control intervention.

Through the training of OHS or general medical practitioners and by computerised self-help interventions the investigators may have better chance to make CBT-I more accessible to a larger number of insomniacs also with different types of working hours. Additionally, it may be possible to decrease chronic insomnia and unfavourably consequences of insomnia to the health and performance capacity in shift workers.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Insomnia (F51.0)
* Difficulty initiating and/or maintaining sleep for ≥ 30 minutes and/or the use of sleep promoting medicine on three or more nights per week for at least 3 months
* Motivation to treat insomnia with non-pharmacological methods
* Full-time shift work (at least 10 % of shifts are morning, evening and/or night shifts)
* Fluent Finnish (due to interventions)

Exclusion Criteria:

* Non-assessed or untreated somatic or mental illness which may explain insomnia
* Planned changes in the work (for example retirement)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes over the measurement points in Insomnia Severity Index (ISI) | Baseline, immediately after intervention and 3-, 6-, 12- and 24-month follow-ups

SECONDARY OUTCOMES:
Changes over the measurement points in sleep diary | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in Sleep Hygiene Practice Scale | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in actigraphy | Baseline, immediately after intervention and 6-month follow-up
Changes over the measurement points in Shirom-Melamed Burnout Measure (SMBM) | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in Generalized Anxiety Disorder (GAD-7) | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in Beck Depression Inventory | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in a single-item measure of stress symptoms | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16) | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in Penn State Worry Questionnaire (PSWQ) | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in Sense of Coherence | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in RAND SF-36 | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
  Finnish version of the RAND 36 item Health Survey
Changes over the measurement points in Work Ability Index | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in Own recovery evaluation | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in Work Cognitive Failure Scale (WCFS) | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in computerized cognitive performance tests | Baseline, immediately after intervention and 6-, 12- and 24-month follow-ups
Changes over the measurement points in blood samples | Baseline and 6-month follow-up
  Genetic analyses

OTHER OUTCOMES:
Short Five (S5) Personality traits (NEO-PRI-R) | Baseline
  Personality traits (Big Five facets)

CONTACTS AND LOCATIONS:
Locations (5):
- Finland (5):
  - City of Helsinki, Occupational Health Centre, Helsinki, Uusimaa
  - Aava Medical Centre, Helsinki
  - Finnair Health Services, Helsinki
  - City of Turku, Occupational Health Centre, Turku
  - Fazer Health Services, Vantaa

REFERENCES:
- [Derived] Jarnefelt H, Harma M, Sallinen M, Virkkala J, Paajanen T, Martimo KP, Hublin C. Cognitive behavioural therapy interventions for insomnia among shift workers: RCT in an occupational health setting. Int Arch Occup Environ Health. 2020 Jul;93(5):535-550. doi: 10.1007/s00420-019-01504-6. Epub 2019 Dec 18. PMID 31853633